CLINICAL TRIAL: NCT00711035
Title: Most Closely HLA Matched Allogeneic Virus Specific Cytotoxic T-Lymphocytes (CTL) to Treat Persistent Reactivation Or Infection With Adenovirus, CMV and EBV After Hemopoietic Stem Cell Transplantation (HSCT)
Brief Title: Most Closely HLA Matched Allogeneic Virus Specific Cytotoxic T-Lymphocytes (CTL)
Acronym: CHALLAH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); M.D. Anderson Cancer Center (Other); National Marrow Donor Program (Other); The Emmes Company, LLC (Industry); Duke University (Other); Beth Israel Deaconess Medical Center (Other); Children's Hospital Los Angeles (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston Children's Hospital (Other); University of Miami (Other); Hackensack Meridian Health (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Helen Heslop, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22994-CHALLAH; CHALLAH; U54HL081007 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-07-08 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Adenovirus Infection; EBV Infection
Keywords: CMV; Adenovirus; EBV; non-myeloablative transplants; Prior allogeneic hematopoietic stem cell transplant
MeSH Terms: conditions — Adenoviridae Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trivirus Specific CTLs for EBV, CMV and Adenovirus Infection (Experimental): If a patient has a partial response they are eligible to receive up to 4 additional doses at biweekly intervals. These doses would come from the original infused line if sufficient vials were available but may come from another line if there are insufficient cells in the original line.
  Interventions: Biological: Trivirus Specific CTLs for EBV, CMV and Adenovirus Infection

INTERVENTIONS:
Biological: Trivirus Specific CTLs for EBV, CMV and Adenovirus Infection — Follow-up Assessments: The timing of follow-up visits is based on the date of CTL infusion. If a patient has multiple CTL doses the schedule resets again at the beginning so follow up relates to the last CTL dose.
  Follow up will occur at 7 days, 14 days, 21 days, 28 days, 42 days, 90 days, 180 days, and 365 days post enrollment.

SUMMARY:
This trial is designed to evaluate the feasibility, safety and efficacy of most closely HLA-matched multivirus specific CTL lines (CHM-CTLs) in HSCT patients with EBV, CMV or adenovirus infections that are persistent despite standard therapy.

The primary objective of the study is to assess safety and feasibility of administering CTLs. Survival data will be collected by asking the transplant center to submit the routine Transplant Essential Data form that is sent to the Stem Cell Transplant Outcomes Database at 100 days and 1 year and includes data on survival status and other outcome measures.

DETAILED DESCRIPTION:
Patients may be screened for study entry when they have persistent disease despite standard therapy as defined in the inclusion criteria. At that stage a search will be done of the available lines. Lines were generated from HSCT donors who consented to the use of CTLs not required for their recipient for research or from normal donors. All donors were screened and deemed to be eligible as transplant donors. We will also manufacture additional lines with the goal of covering common HLA types and will consult with the NMDP to determine what HLA types would be desirable. Additional donors will be screened by a transplant donor center physician and must be deemed eligible before a line can be manufactured.

CTL Lines: We will use trivirus specific CTL lines generated as described previously. Generation of trivirus-specific CTL lines requires the generation of several different components from PBMC. The CTL line will be derived from donor peripheral blood T cells, by multiple stimulations with antigen-presenting cells (APCs) presenting CMV, EBV and adenovirus antigens and expansion with interleukin-2 (IL-2). The APCs used to stimulate and expand the CMV-specific T cells will be derived from patient mononuclear cells and B lymphocytes.

To initiate the trivirus-specific CTL line, PBMC will be transduced with an adenovirus vector (Ad5f35-pp65) expressing the immunodominant antigen of CMV, pp65. The monocyte fraction of PBMC expressed and presented CMV-pp65 peptide epitopes to the CMV-specific T cell fraction of the PBMC, while the virion proteins from the adenovirus vector were processed and presented to the adenovirus-specific T cell fraction.

To expand trivirus -specific T cells we used EBV-transformed B lymphoblastoid cell lines (EBV-LCLs) transduced with Ad5f35-pp65. This transduction allows the EBV-LCLs to present CMV-pp65 and adenovirus virion peptides to the T cells as well as endogenously expressed EBV antigens.

EBV-LCLs are derived from PBMC-B lymphocytes by infection with a clinical grade, laboratory strain of Epstein-Barr virus (EBV). About 5 x 10^6 PBMC, or 5 to 10 mLs of blood is required to generate the EBV-LCL

At the end of the CTL culture period, the frequency of T cells specific for each virus were determined using tetramer reagents if available. To test the functional antigen specificity of the CTL we will use overlapping peptide libraries for pp65 and adenovirus hexon and autologous and allogeneic LCLs in Elispot assays and we will perform cytotoxicity assays using unmodified PHA blasts and LCLs untransduced or transduced with Adhexon and CMVpp65 pepmix OR LCL transduced with Ad5f35-null and Ad5f35-pp65. Some lines will have aliquots sent for further characterization to the NIH where Drs Melenhorst and Barrett are developing assays to predict alloreactivity where they examine virus antigen-specific T cells using an extensive panel of activated T cells as antigen presenting cells (T-APC). These lines will be labeled with component number only and will not have subject identifiers.

The CTL lines will also be checked for identity, phenotype and sterility, and cryopreserved prior to administration according to SOP. Release criteria for administering the CTL to patients include viability >70%, negative culture for bacteria and fungi for at least 7 days, endotoxin testing less than or equal to 5EU/ml, negative result for Mycoplasma, <2% CD19 positive B cells, <2% CD14 positive monocytes (or <2% CD83 positive cells if Dendritic cells were used as stimulators) and HLA identity.

No Matched CTL Line Available: If no matched line is available the patient will be registered so that the feasibility of the approach can be assessed and the eventual outcome will also be collected.

CTL Line Available but Patient Status Changes: Patients clinical course that changes between screening and infusion will not be given the CTL and will be followed for eventual outcome.

Survival data will be collected by asking the transplant center to submit the routine Transplant Essential Data form that is sent to the Stem Cell Transplant Outcomes Database at 100 days and 1 year and includes data on survival status and other outcome measures.

Criteria for Selection of CTL Line: In general the line matching at the highest number of HLA loci will be selected. Matching at the allele level will be preferred but antigen level will be accepted or HLA-A and HLA-B. However consideration will also be given to the type of infection and activity of the line against that virus. For example for a patient with adenovirus infection a line that matches at 2 loci but that has recognition of adenovirus mediated through those antigens would be preferable to a line matched at 3 loci but with no demonstrated activity against adenovirus. The protocol chair will discuss each case with the principal investigators at each center to determine the optimal CTL line for each patient. If more than one line matches and there are insufficient cells to cover additional infusions a second CTL line will be reserved in the event that additional infusions are warranted. Patients with a partial response are eligible to receive an additional dose.

Premedications: Patients will be premedicated with Benadryl 1mg/kg (max 50 mg) IV and Tylenol 10 mg/kg (max 650 mg) PO.

Patients will be monitored according to institutional standards for administration of blood products and at a minimum will be monitored according to below: • Patients should remain in the clinic for at least one hour • Patients should remain on continuous pulse oximetry for at least 30 minutes • Vital signs should be monitored at the end of infusion then at 30 and 60 minutes

Supportive Care: Patients will receive supportive care for acute or chronic toxicity, including blood components or antibiotics, and other intervention as appropriate.

If a patient has a partial response they are eligible to receive up to 4 additional doses at a minimum 2 week intervals and if they meet the eligibility criteria for subsequent lines. These doses would come from the original infused line if sufficient vials were available but may come from another line if there are insufficient cells in the original line.

Follow-up Assessments: The timing of follow-up visits is based on the date of CTL infusion. If a patient has multiple CTL doses the schedule resets again at the beginning so follow up relates to the last CTL dose.

Follow up will occur at 7 days, 14 days, 21 days, 28 days, 42 days, 90 days, 180 days, and 365 days (+/- 2 days up to Week 8, and +/- 14 days for Days 90, 120, and +/- 28 days for 6 and 12 months, post-enrollment..)

The following assessments are considered standard-of-care unless identified below by " * ":

Pre-Infusion: 1. History and physical exam including height and weight 2. Viral loads for EBV, adenovirus, CMV 3. Biopsy disease site, if appropriate 4. Imaging studies, if appropriate 5. Complete acute GVHD staging and grading information including assessments of rash, diarrhea, nausea/vomiting, weight and liver function tests 6. CBC with differential, platelet count 7. Liver function tests (bilirubin, alkaline phosphatase, AST, ALT) plus creatinine 8. Tacrolimus/cyclosporine level 9. * Samples for laboratory studies

Post-Infusion: 1. Viral loads for CMV, EBV, adenovirus weekly at 1, 2, 3, 4 and 6 weeks and 3, 6 and 12 months. 2. Complete acute GVHD staging and grading information including assessments of rash, diarrhea, nausea/vomiting, weight and liver function tests weekly until Day 45 3. Chronic GVHD evaluation (if present) 3, 6, 9, and 12 months 4. CBC with differential and platelet count at 1, 2, 3, 4, and 6 weeks. 5. Infusion related toxicities within 24 hours and toxicity evaluation weekly until Day 30 and acute GVHD until Day 45 6. Steroid dose weekly until Day 42, and 3, 6 and 9 months 7. * Samples for laboratory studies on Days 0, 14, 28 and 90 8. Infections through Day 42 and at 3, 6 and 12 months

Ancillary laboratory studies will include: 1) Assessment of virus-specific immunity based on CTL levels as measured by ELISPOT assays or tetramer assays. 2) Persistence of infused T cells based on PCR for non-shared antigen

Reporting Patient Deaths: The Recipient Death Information must be entered into the web-based data entry system within 24 hours of knowledge of a patient's death. If the cause of death is unknown at that time, it need not be recorded at that time. However, once the cause of death is determined, the form must be updated.

Donor Evaluation: - Complete history and physical examination - CBC, platelets, differential - Total protein, albumin, total bilirubin, alkaline phosphatase, ALT, AST, - HIV-1 antibody, HIV-2 antibody, HIV NAT, HTLV-1/2 antibodies, HBsantigen, HBc antibody, HCV NAT, CMV antibody, RPR, West Nile virus NAT, and Chagas testing - ABO and Rh typing - When the evaluation is complete, the Transplant Physician will note in the recipient's and donor's medical records that the tests have been evaluated, and the donor is acceptable.

ELIGIBILITY:
INCLUSION CRITERIA:

Pts will be eligible following any type of allogeneic transplant if they have CMV, adenovirus or EBV infection persistent to standard therapy (as defined below).

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow, peripheral blood stem cells or single or double cord blood within 18 months.
2. CMV, adenovirus or EBV infection persistent despite standard therapy

   1. For CMV infection: i.Pts with CMV disease: defined as the demonstration of CMV by biopsy specimen from visceral sites (by culture or histology) or the detection of CMV by culture or direct fluorescent antibody stain in bronchoalveolar lavage fluid in the presence of new or changing pulmonary infiltrates OR ii. Failure of antiviral therapy: defined as the continued presence of pp65 antigenemia (>1+ cell/100,000 cells) or DNAemia (as defined by reference lab performing PCR assay but usually >400 copies/ml) after at least 7 days of antiviral therapy OR iii. Relapse after antiviral therapy defined as recurrence of either pp65 antigenemia or DNAemia after at least 2 weeks of antiviral therapy iv. For CMV infection, standard therapy is defined as 7 days therapy with Ganciclovir, Foscarnet or Cidofovir for patients with disease or recurrence after 14 days therapy
   2. For EBV infection: i. EBV infection is defined as: 1. Biopsy proven lymphoma with EBV genomes detected in tumor cells by immunocytochemistry or in situ PCR OR 2. Or clinical or imaging findings consistent with EBV lymphoma and elevated EBV viral load in peripheral blood. ii. For EBV infection, standard therapy is defined as rituximab given at 375mg/m^2 in patients for 1-4 doses with a CD20+ve tumor iii. Failure is defined as: 1. There was an increase or less than 50% response at sites of disease for EBV lymphoma OR 2. There was a rise or a fall of less than 50% in EBV viral load in peripheral blood or any site of disease
   3. For adenovirus infection or disease: i. Adenovirus infection is defined as the presence of adenoviral positivity as detected by PCR, DAA or culture from ONE site such as stool, blood, urine, or nasopharynx OR ii. Adenovirus disease will be defined as the presence of adenoviral positivity as detected by culture from two or more sites such as stool or blood or urine or nasopharynx iii. Standard therapy is defined as 7 days therapy with Cidofovir (if renal function permits this agent to be given) iv. Failure is defined as a rise or a fall of less than 50% in viral load in peripheral blood or any site of disease as measured by PCR or any other quantitative assay)
3. Pts with multiple CMV, EBV or Adenovirus infections are eligible given that each infection is persistent despite standard therapy as defined above. Patients with multiple infections with one persistent infection and one controlled infection are eligible to enroll.
4. Clinical status at enrollment to allow tapering of steroids to less than 0.5 mg/kg/day prednisone.
5. Written informed consent from patient, parent or guardian.
6. Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).

The informed consent process will begin at recognition of subject eligibility and consent will be obtained per institutional practices before study therapy is initiated. Subjects will initially sign a screening consent to enable a search to be made for a line. If a line is available they will sign the treatment consent.

Up to 4 additional doses can be administered if a partial response is obtained and patient meets eligibility criteria for subsequent infusions. The minimum interval between subsequent infusions is 2 weeks.

Donors will be eligible if they meet eligibility criteria for blood donors on history and exam by a transplant donor physician and have negative infectious diseases testing.

EXCLUSION CRITERIA:

For initial CTL and subsequent infusions:

1. Patients receiving ATG, or Campath or other immunosuppressive monoclonal antibodies within 28 days of screening for enrollment.
2. Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.

   Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
3. Patients who have received donor lymphocyte infusion (DLI) within 28 days.
4. Patients with active acute GVHD grades II-IV.
5. Active and uncontrolled relapse of malignancy

Donors will be ineligible if they do not meet eligibility criteria for blood donors on the donor questionnaire or have positive infectious diseases testing on any of the tests outlined in the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The primary purpose of the study is to assess the safety of administering CHM-CTLs in transplant patients with EBV, CMV, or adenovirus infection. We have elected to use a dose of 2 x 10^7 CHM-CTLs/m2. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (8):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Miami, Coral Gables, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University, Bergen County, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Leen AM, Bollard CM, Mendizabal AM, Shpall EJ, Szabolcs P, Antin JH, Kapoor N, Pai SY, Rowley SD, Kebriaei P, Dey BR, Grilley BJ, Gee AP, Brenner MK, Rooney CM, Heslop HE. Multicenter study of banked third-party virus-specific T cells to treat severe viral infections after hematopoietic stem cell transplantation. Blood. 2013 Jun 27;121(26):5113-23. doi: 10.1182/blood-2013-02-486324. Epub 2013 Apr 22. PMID 23610374